CLINICAL TRIAL: NCT03050892
Title: Impact of Donor and Recipient ST2 / IL-33 Pathway on Recipient Survival and Acute Rejection After Heart Transplantation
Brief Title: Impact of Donor and Recipient ST2 / IL-33 Pathway After Heart Transplantation
Acronym: ISIDORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Antonella Galeone, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC-1421-16-01
Record Dates: First submitted 2017-02-05; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Heart Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the association between donor soluble protein ST2 (sST2) serum levels and 30-day recipient mortality in order to improve graft screening.

DETAILED DESCRIPTION:
Soluble protein sST2 has recently become a prognostic biomarker in the context of acute myocardial infarction and chronic heart failure, and recent studies also show that sST2 is involved in acute rejection of the cardiac graft in recipients. Experimental studies confirm that the ST2 / IL-33 pathway is involved in the process leading to cardiac transplant rejection in animals. In particular, administration of IL-33 would have a positive effect on pre-clinical cardiac graft survival. No study have looked at the level of ST2 / IL-33 of the donor, with the purpose that it might reflect the condition of the transplanted heart and its initial level of Immune tolerance and maybe predict the risk of subsequent dysfunction.

In this non-interventional study, several blood samples will be taken on donors before organ procurement and on recipients prior to grafting, on day 7 and at the time of each myocardial biopsy (approximately 16 myocardial biopsies the first year). Serum level of sST2 and IL-33 will then be determined according to the ELISA method on each blood sample.

Fifty consecutive couple donors/ recipients will be included in the study. This number of subjects is calculated to detect a doubling of the donor sST2 level between the two recipient groups with 30-day mortality and without mortality (potency: 90%, alpha risk: 0.05, bilateral).

ELIGIBILITY:
Inclusion Criteria:

* Consenting recipients
* Consenting donors to organ/tissue donation for the purpose of scientific research

Exclusion Criteria:

* Non consenting recipients
* Non consenting donors to organ/tissue donation for the purpose of scientific research
* Multi-organ transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart donors and heart recipients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-03-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 30 days
  Compare mean donor sST2 serum levels in recipients who died at 30 days versus mean donor sST2 serum levels in recipients who survived at 30 days.

SECONDARY OUTCOMES:
Survival and Rejection and IL-33 | 1 year
  * Compare mean donor IL-33 serum levels in recipients with 30 days events (mortality and graft dysfunction) versus mean donor IL-33 serum levels in recipients without 30 days events.
  * Compare mean donor IL-33 serum levels in recipients with one year events (mortality and / or graft dysfunction) versus mean donor IL-33 serum level in recipients without events.
  * Compare mean IL-33 serum levels of recipients with events (mortality and / or graft dysfunction) at 30 days and 1 year versus mean IL- 33 serum levels of the recipients who had no events at 30 days and 1 year.
  * Compare the mean donor and recipient IL-33 serum levels in recipients with acute graft rejection versus mean donor and recipient IL-33 serum levels in recipients who did not have an acute rejection of the graft during the first year.
Survival and Rejection and sST2 | 1 year
  * Compare mean donor sST2 serum levels in recipients with one year events (mortality and / or graft dysfunction) versus mean donor sST2 serum level in recipients without events.
  * Compare mean sST2 serum levels of recipients with events (mortality and / or graft dysfunction) at 30 days and 1 year versus mean sST2 serum levels of the recipients who had no events at 30 days and 1 year.
  * Compare the mean donor and recipient sST2 serum levels in recipients with acute graft rejection versus mean donor and recipient sST2 serum levels in recipients who did not have an acute rejection of the graft during the first year.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Cardiac Institute, Groupe Hospitalier La Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No